CLINICAL TRIAL: NCT01769976
Title: Effects of Periodic Fasting Versus Daily Energy Restriction on Metabolic Health
Acronym: PREFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, A/Prof Leonie Heilbronn, Associate Professor, University of Adelaide
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APP1023401
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Daily energy restriction (Experimental): 25% reduction in daily energy intake
  Interventions: Other: Energy restriction
- Energy balance diet (Active Comparator): Diet provides 100% of energy requirements and is designed to achieve weight stability
  Interventions: Other: Energy balance diet
- Periodic fasting with weight loss (Experimental): Fast 3 days per week, and consume 1.5 times usual amount of food on other days
  Interventions: Other: Periodic fasting; Other: Energy restriction
- Periodic fasting without weight loss (Experimental): Fast 3 days per week, and consume double usual amount of food on other days
  Interventions: Other: Periodic fasting; Other: Energy balance diet

INTERVENTIONS:
Other: Periodic fasting
  Arms: Periodic fasting with weight loss; Periodic fasting without weight loss
Other: Energy restriction
  Arms: Daily energy restriction; Periodic fasting with weight loss
Other: Energy balance diet
  Arms: Energy balance diet; Periodic fasting without weight loss

SUMMARY:
The aim of this study is to examine whether periodic fasting improves markers of diabetes risk and cardiovascular health, and will compare this to the effects observed with daily dieting by energy restriction, and also with no change in energy intake.

It is hypothesized that periodic fasting, with or without weight loss, will be as effective as daily energy restriction to improve markers of metabolic health and energy metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25 and 42 kg/m2
* weight stable (<5% fluctuation in body weight for the 6 months prior to study entry)

Exclusion Criteria:

* history of cardiovascular disease, diabetes, major psychiatric disorders, and eating disorders
* use of prescribed or non-prescribed medications with may affect energy metabolism, gastrointestinal function, body weight, or appetite
* recent weight changes in 3 months prior to study entry
* uncontrolled asthma, current fever, upper respiratory infections
* individuals who regularly perform high intensity exercise (>2 sessions per week)
* pregnancy, lactation (breast feeding), women who are planning to become pregnant
* current intake of >140g of alcohol per week
* current smoker of cigarettes/cigars/marijuana
* current intake of any illicit substance
* experience claustrophobia in confined spaces
* has donated blood within the past 3 months
* unable to comprehend the study protocol
* experiences migraines

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 8 weeks
  assessed by hyperinsulinemic euglycemic clamp

SECONDARY OUTCOMES:
Plasma hormones and adipokines | 8 weeks
Cognitive function, hunger, and mood | 8 weeks
Oxidative stress, stress resistance, and lipid metabolism | 8 weeks
Energy expenditure | 8 weeks
  resting energy expenditure, and total daily energy expenditure

CONTACTS AND LOCATIONS:
Overall Officials: Leonie Heilbronn, Principal Investigator — University of Adelaide
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- [Derived] Hutchison AT, Liu B, Wood RE, Vincent AD, Thompson CH, O'Callaghan NJ, Wittert GA, Heilbronn LK. Effects of Intermittent Versus Continuous Energy Intakes on Insulin Sensitivity and Metabolic Risk in Women with Overweight. Obesity (Silver Spring). 2019 Jan;27(1):50-58. doi: 10.1002/oby.22345. PMID 30569640
- [Derived] Chen M, Liu B, Wilkinson D, Hutchison AT, Thompson CH, Wittert GA, Heilbronn LK. Selenoprotein P is elevated in individuals with obesity, but is not independently associated with insulin resistance. Obes Res Clin Pract. 2017 Mar-Apr;11(2):227-232. doi: 10.1016/j.orcp.2016.07.004. Epub 2016 Aug 11. PMID 27524654